CLINICAL TRIAL: NCT03344380
Title: Identification of Genetic Polymorphism Related to Acute Kidney Injury After Liver Transplantation Through Genome-wide Association Study (GWAS) in Korean Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0888
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: The Recipients Undergoing Liver Transplantation
Keywords: Gene polymorphism; acute kidney injury; liver transplantation
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood obtained from enrolled patients before surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: Adult patients undergoing liver transplantation will be included and followed up during the first 72 hours post-liver transplantation in order to confirm the development of acute kidney injury. The patients will be divided into two groups (AKI group vs. non-AKI group) according to the development of acute kidney injury. The GWAS will be performed with the blood obtained from enrolled patients.
- Retrospective cohort: In previous study performed in adult patients undergoing liver transplantation (NCT02489474, 4-2015-0411), we enrolled patients and collected data regarding the development of acute kidney injury during the first 72 hours post-liver transplantation. Among these patients enrolled in this previous study, only patients who agreed to additional use of the blood sample for research purposes will be included in the present study. The GWAS will be performed with the blood obtained from enrolled patients.

SUMMARY:
Some of the liver transplantation recipients experience postoperative acute kidney injury due to various causes including genetic factors. Prevention of postoperative acute kidney injury is essential for postoperative care in liver transplantation recipients. The aim of this study is to investigate the relationship between gene polymorphisms and the occurrence of acute kidney injury after liver transplantation by performing genome-wide association study (GWAS).

ELIGIBILITY:
Inclusion Criteria:

1) adult patients scheduled for liver transplantation

Exclusion Criteria:

1. Patients on dialysis
2. patients not able to read, or understand the consent form
3. ethnicity, other than asian
4. patients refusal

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury after liver transplantation | Participants will be followed up during the first 72 hours post-liver transplantation in order to confirm the development of acute kidney injury.
  The development of acute kidney injury is defined by the following definition: 50% increase in SCr from the baseline (preoperative value) or a 0.3 mg/dl increase from baseline within 48 h without urine output. The development of acute kidney injury after liver transplantation could correlate with gene polymorphisms, which have been known to be associated with postoperative acute kidney injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea